CLINICAL TRIAL: NCT07008027
Title: Real World Asparaginase Therapy Toxicity
Status: Not yet recruiting | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: REWASPY
Record Dates: First submitted 2025-05-28; First posted 2025-06-06 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Drug Toxicity
Keywords: Asparaginase drugs; Toxicity; Acute lymphoblastic leukemia; Acute lymphoblastic lymphoma; Mixed phenotype acute leukemia
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Biphenotypic, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-protocol therapy /standard of care therapy: Participants receiving non -protocol standard if care (SOC) treatment.
- SJALL23T (NCT06390319) protocol therapy: Participants receiving protocol therapy on SJALL23T and not receiving investigational drug.

SUMMARY:
This research study is being done to learn more about the short term and long term side effects of treatment with asparaginase drugs, which are commonly used in acute lymphoblastic leukemia (ALL) or acute lymphoblastic lymphoma (LLy) therapy.

DETAILED DESCRIPTION:
Primary Objective

* To estimate the rate of high-grade toxicities which occur during therapy for acute lymphoblastic leukemia/ lymphoma in patients receiving asparaginase-containing standard of care therapy.

This study will involve the collection of data about the participants ALL/LLy, treatment, side effects of treatment and leukemia/ lymphoma's response to treatment. Data collected on other research studies participants are enrolled on will also be used for this research study.

Blood samples will be collected and liver fibroscans (liver ultrasounds) will be done at different time points while the participant is receiving treatment for ALL/LLy. The time points will depend on what treatment they receive and will correspond to days on their treatment roadmap.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of acute lymphoblastic leukemia, lymphoblastic lymphoma, or mixed phenotype acute leukemia
* Enrolled on INITIALL and no more than 10 days after initiation of post-INITIALL therapy
* Post-INITIALL therapy is:

  * Standard of Care (SOC)/Non Protocol Treatment Plan (NPTP) as per Total therapy or
  * SJALL23T and not scheduled to receive venetoclax

Exclusion Criteria:

* Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants meeting the Eligibility Criteria.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2030-07 (Estimated); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Probability of developing CTCAE grade 3+ (3, 4, 5) or 4+ (4, 5) toxicities during standard of care (SOC) therapy | Approximately 2½ to 3 years
  The overall probability of on-therapy grade 3+ or 4+ toxicity will be estimated by the sample proportion along with the Normal approximation (Z-statistic) based 95% confidence interval.
Probability of developing CTCAE grade 3+ (3, 4, 5) or 4+ (4, 5) toxicities SJALL23T therapy | Approximately 2½ to 3 years
  The overall probability of on-therapy grade 3+ or 4+ toxicity will be estimated by the sample proportion along with the Normal approximation (Z-statistic) based 95% confidence interval.
Cumulative incidence (CIN) of the grade 3+ or 4+ toxicities throughout SOC therapy | Approximately 2½ to 3 years
  Cumulative incidence (CIN) of the grade 3+ or 4+ toxicities throughout therapy will be estimated using the Kalbafleisch-Prentice method.
Cumulative incidence (CIN) of the grade 3+ or 4+ toxicities throughout SJALL23T therapy | Approximately 2½ to 3 years
  Cumulative incidence (CIN) of the grade 3+ or 4+ toxicities throughout therapy will be estimated using the Kalbafleisch-Prentice method.
Probabilities of grade 3+ or 4+ toxicities each phase of SOC treatment | Approximately 2½ to 3 years
  Probabilities of grade 3+ or 4+ toxicities will be estimated for each treatment phase by sample proportions accompanied by the Z-statistic 95% confidence intervals.
Probabilities of grade 3+ or 4+ toxicities each phase of SJALL23Ttreatment | Approximately 2½ to 3 years
  Probabilities of grade 3+ or 4+ toxicities will be estimated for each treatment phase by sample proportions accompanied by the Z-statistic 95% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Seth E. Karol, MD, MSCI, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols